CLINICAL TRIAL: NCT03293095
Title: Functional Task Kinematic in Patient With Musculoskeletal Pathology.
Brief Title: Functional Task Kinematic in Musculoskeletal Pathology.
Status: Completed | Type: Observational
Sponsor: University of Malaga (Other)
Collaborators: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Dr. Antonio I Cuesta-Vargas, PhD, University of Malaga
Other Study IDs: iBAFI01
Record Dates: First submitted 2017-09-21; First posted 2017-09-26 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2019-07

CONDITIONS: Musculoskeletal Disease
Keywords: musculoskeletal pathology; motion sensor; motion capture; functional task; biomarker
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute musculoskeletal pathology patients: Musculoskeletal pathology patients that they will perform functional tasks measuring with motion sensors and motion capture.
  Interventions: Procedure: Standard Care
- Match control: Healthy people of the same age as the acute musculoskeletal pathology subjects. They will perform functional tasks measuring with motion sensors and motion capture.
  Interventions: Procedure: Standard Care

INTERVENTIONS:
Procedure: Standard Care — The guidelines for the management according to the musculoskeletal disorder in primary care will be the treatment guidelines for the Standard Care.

SUMMARY:
The aim of this project is to create references values to patients with musculoskeletal pathology using functional tasks and measuring with a smartphone and video imaging (3D motion capture cameras).

DETAILED DESCRIPTION:
Musculoskeletal pathologies can affect bones, muscles, joints and other structures related to this system. These disorders are extremely common and can have an origin from autoimmune, inflammatory, traumatic, etc. The risk of developing this pathologies increases with age.

The diagnosis could delayed by lack of information, expensive assessment or difficult execution.

Currently, you can use a Smartphone to get the same information as sensors. In addition to Smartphone, 3D motion capture systems with a camera have been frequently used to analyse kinematics and are being integrated as a rehabilitation tool in patients. The use of Smartphones and 3D motion capture cameras would help to find fast and cheap assessment methods for professionals.

ELIGIBILITY:
Inclusion Criteria:

* Persons with diagnosis of musculoskeletal pathology.
* Age between 20-65 años.
* Subjects able to get up from the chair at least 5 times.
* Be able to complete questionnaires and perform functional tasks.

Exclusion Criteria:

* Subjects who are participating in a study with an experimental treatment.
* Severe cardiovascular disease.
* Being pregnant, in case of women.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients treat in general care or diagnosed by a specialist.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Kinematic analysis by motion sensor | 1 hour
  A smartphone will pick up positioning, motion and acceleration information from the subject
Kinematic analysis by 3D motion capture | 1 hour
  The camera will perform a motion capture of the functional task. This system will calculate the displacement and the time of the functional task
Responsiveness | 1 hour
  The Responsiveness Box of COSMIN checklist will be used to determinate the response to change of the Smartphone and the 3D cameras. All possible items will be followed.

SECONDARY OUTCOMES:
Quality of life questionnaire: EuroQoL 5D | 1 hour
  standardized instrument for use as a measure of health outcome

CONTACTS AND LOCATIONS:
Overall Officials: Antonio I Cuesta-Vargas, PhD, Principal Investigator — University of Malaga
Locations (1):
- Malaga, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kilic G, Kilic E, Ozgocmen S. Relationship between psychiatric status, self-reported outcome measures, and clinical parameters in axial spondyloarthritis. Medicine (Baltimore). 2014 Dec;93(29):e337. doi: 10.1097/MD.0000000000000337. PMID 25546683
- [Background] Galan-Mercant A, Baron-Lopez FJ, Labajos-Manzanares MT, Cuesta-Vargas AI. Reliability and criterion-related validity with a smartphone used in timed-up-and-go test. Biomed Eng Online. 2014 Dec 2;13:156. doi: 10.1186/1475-925X-13-156. PMID 25440533
- [Background] Moreno FA, Merchan-Baeza JA, Gonzalez-Sanchez M, Gonzalez-Jimenez J, Cuesta-Vargas AI. Experimental Validation of Depth Cameras for the Parameterization of Functional Balance of Patients in Clinical Tests. Sensors (Basel). 2017 Feb 22;17(2):424. doi: 10.3390/s17020424. PMID 28241455
- [Background] van Weely SF, van Denderen CJ, van der Horst-Bruinsma IE, Nurmohamed MT, Dijkmans BA, Dekker J, Steultjens MP. Reproducibility of performance measures of physical function based on the BASFI, in ankylosing spondylitis. Rheumatology (Oxford). 2009 Oct;48(10):1254-60. doi: 10.1093/rheumatology/kep190. Epub 2009 Jul 28. PMID 19638455
- [Background] Fritz JM, Piva SR. Physical impairment index: reliability, validity, and responsiveness in patients with acute low back pain. Spine (Phila Pa 1976). 2003 Jun 1;28(11):1189-94. doi: 10.1097/01.BRS.0000067270.50897.DB. PMID 12782991
- [Background] van Tulder M, Becker A, Bekkering T, Breen A, del Real MT, Hutchinson A, Koes B, Laerum E, Malmivaara A; COST B13 Working Group on Guidelines for the Management of Acute Low Back Pain in Primary Care. Chapter 3. European guidelines for the management of acute nonspecific low back pain in primary care. Eur Spine J. 2006 Mar;15 Suppl 2(Suppl 2):S169-91. doi: 10.1007/s00586-006-1071-2. No abstract available. PMID 16550447
- [Background] Mokkink LB, Terwee CB, Patrick DL, Alonso J, Stratford PW, Knol DL, Bouter LM, de Vet HC. The COSMIN checklist for assessing the methodological quality of studies on measurement properties of health status measurement instruments: an international Delphi study. Qual Life Res. 2010 May;19(4):539-49. doi: 10.1007/s11136-010-9606-8. Epub 2010 Feb 19. PMID 20169472
- [Background] Dankaerts W, O'Sullivan P. The validity of O'Sullivan's classification system (CS) for a sub-group of NS-CLBP with motor control impairment (MCI): overview of a series of studies and review of the literature. Man Ther. 2011 Feb;16(1):9-14. doi: 10.1016/j.math.2010.10.006. Epub 2010 Nov 20. PMID 21094624
- [Background] Myers AM, Holliday PJ, Harvey KA, Hutchinson KS. Functional performance measures: are they superior to self-assessments? J Gerontol. 1993 Sep;48(5):M196-206. doi: 10.1093/geronj/48.5.m196. PMID 8366262
- [Background] Roldan-Jimenez C, Bennett P, Cuesta-Vargas AI. Muscular Activity and Fatigue in Lower-Limb and Trunk Muscles during Different Sit-To-Stand Tests. PLoS One. 2015 Oct 27;10(10):e0141675. doi: 10.1371/journal.pone.0141675. eCollection 2015. PMID 26506612
- [Derived] Trinidad-Fernandez M, Beckwee D, Cuesta-Vargas A, Gonzalez-Sanchez M, Moreno FA, Gonzalez-Jimenez J, Joos E, Vaes P. Differences in movement limitations in different low back pain severity in functional tests using an RGB-D camera. J Biomech. 2021 Feb 12;116:110212. doi: 10.1016/j.jbiomech.2020.110212. Epub 2020 Dec 27. PMID 33401131
- [Derived] Trinidad-Fernandez M, Beckwee D, Cuesta-Vargas A, Gonzalez-Sanchez M, Moreno FA, Gonzalez-Jimenez J, Joos E, Vaes P. Validation, Reliability, and Responsiveness Outcomes Of Kinematic Assessment With An RGB-D Camera To Analyze Movement In Subacute And Chronic Low Back Pain. Sensors (Basel). 2020 Jan 27;20(3):689. doi: 10.3390/s20030689. PMID 32012763